CLINICAL TRIAL: NCT06466915
Title: Comparison of the Use of Propofol and Nasal Dexmedetomidine in the Management of Agitation and Delirium in Patients Undergoing Dental Procedures
Brief Title: Propofol vs. Nasal Dexmedetomidine in Pediatric Agitation and Delirium
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Baskent University Ankara Hospital (Other)
Responsible Party: Principal Investigator, Ahmed Uslu, MD, Research assistant, Baskent University Ankara Hospital
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: PedSed
Record Dates: First submitted 2024-06-14; First posted 2024-06-20 (Actual); Last update posted 2025-01-17 (Actual); Status verified 2025-01

CONDITIONS: Comparison of the Effects of Propofol and Nasal Dexmedetomidine
MeSH Terms: interventions — Dexmedetomidine; Propofol

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No | US Export: Yes

ARMS (3):
- Group Dex (Experimental): Group Dex received 1 mcg/kg of dexmedetomidine intra-nasal 10 minutes before the surgical procedure ended.
  Interventions: Drug: Dexmedetomidine
- Group Pofol (Experimental): Group Pofol received 1 mg/kg propofol IV before the extubation.
  Interventions: Drug: Propofol
- Group PoDex (Experimental): Group PoDex received 0.5 mcg/kg of dexmedetomidine intra-nasal 10 minutes before the surgical procedure ended and 0.5 mg/kg propofol IV before the extubation.
  Interventions: Drug: Dexmedetomidine; Drug: Propofol

INTERVENTIONS:
Drug: Dexmedetomidine — Group Dex received 1 mcg/kg of dexmedetomidine intra-nasal 10 minutes before the surgical procedure ended.
  Arms: Group Dex; Group PoDex
Drug: Propofol — Group Pofol received 1 mg/kg propofol IV before the extubation.
  Arms: Group PoDex; Group Pofol

SUMMARY:
Dental pain and anxiety are quite common in pediatric patients. However, due to children's inability to express their fears and lack of knowledge about the procedures to be performed, these symptoms have often been misunderstood and inadequately treated in pediatric settings. Children have consistently experienced high rates of emergence anxiety during the recovery process after general anesthesia. Emergence anxiety can be harmful to the patient, leading to bleeding at the surgical site, displacement of intravenous catheters, parental anxiety, additional care needs, and delays in hospital discharge. Inhalation anesthetics are preferred for pediatric surgeries because they promote faster recovery. However, inhalation anesthetics often lead to a high rate of emergence anxiety, ranging from 25% to 80% depending on the scoring scale used, the child's age, and the type of surgery performed. Additional sedative or analgesic drugs, such as midazolam, dexmedetomidine, or propofol, have been used to prevent emergence anxiety.

Dexmedetomidine is a selective α2-agonist with sedative and analgesic effects, but it can cause mild respiratory depression. Numerous studies have shown that intranasal dexmedetomidine is more effective than other adjunctive drugs. It has been found to be beneficial in reducing emergence anxiety during pediatric anesthesia with minimal blood pressure or respiratory depression. However, although intranasal dexmedetomidine initially has relatively rapid absorption, the absorption process may take longer compared to intravenous administration, implying that the child's hemodynamic status is more stable and a longer effective absorption time may have a clinical advantage in preventing emergence anxiety.

The aim of this study is to compare and investigate the effectiveness of nasal dexmedetomidine and intravenous propofol applications used to reduce agitation in pediatric cases following extubation in clinical practice.

ELIGIBILITY:
Inclusion Criteria:

* ASA 1-2

Exclusion Criteria:

* Cardiac disease,
* Psychiatric disease,
* Coronary artery disease,
* Long-term sedative drug use,
* Pulmonary disease,
* Known allergy to planned drugs

Ages: 1 Year to 8 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 162 (Actual)
Dates: Start 2023-06-01 (Actual); Primary Completion 2024-04-30 (Actual); Study Completion 2024-04-30 (Actual)

PRIMARY OUTCOMES:
Agitation-Delirium | 0, 5, 10, 15, 20, 25, 30. minutes after extubation.
  It will be evaluated with a Pediatric Anesthesia Emergence Delirium Scale.
Behavioral pain assessment | 0, 5, 10, 15, 20, 25, 30. minutes after extubation.
  It will be evaluated with a The Face, Legs, Activity, Cry, and Consolability Scale.

SECONDARY OUTCOMES:
Nausea-vomiting | 0, 5, 10, 15, 20, 25, 30. minutes after extubation.
  It will be evaluated by visual analogue scale.
Rapid recovery | 30 minutes after extubation.
  It will be evaluated with a Modified Aldrete Score.

CONTACTS AND LOCATIONS:
Locations (1):
- Ahmed Uslu, Ankara, Çankaya, Turkey (Türkiye)